CLINICAL TRIAL: NCT06223776
Title: Effects of One Night's Acute Sleep Restrictions on Maximal Strength, Muscle Power, and Strength Endurance in Resistance-trained Women.
Brief Title: Effects of Sleep Restrictions on Maximal Strength, Muscle Power, and Strength Endurance in Resistance-trained Women.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 160/MN/INoS/2023
Record Dates: First submitted 2023-11-10; First posted 2024-01-25 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Sleep Restriction; Sleep
Keywords: acute sleep restriction; early sleep restriction

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal sleep (No Intervention): The night before the experimental session, where participants will follow their habitual sleep-wake routines.
- Sleep restriction (Experimental): The night before the experimental session (with sleep restrictions (SR)), where participants will experience acute sleep restriction the night before the test session (i.e., 3 h of early sleep restriction versus normal sleep).
  Interventions: Procedure: Sleep restriction

INTERVENTIONS:
Procedure: Sleep restriction — Participants will experience a night of acute sleep restriction. During this night, they will sleep 3 hours less than usual.
  Arms: Sleep restriction

SUMMARY:
The study aims to see how acute sleep restriction will affect women resistance trainers. Above all, the investigators will be interested in observing the relationship between shorter sleep and athletic performance, as well as other important aspects, such as their level of motivation to exercise, how much pain participants felt during exercise and how demanding they found exercise. The investigators assume that differences in subjective measures (such as pain levels, motivation and mood) will be most apparent.

DETAILED DESCRIPTION:
Participants would take part in two identical experimental sessions under two sleep conditions:

with sleep restrictions (SR), where will experience acute sleep restriction the night before the test session (i.e., 3 h of early sleep restriction versus normal sleep); with the control condition (CON), where participants will follow their habitual sleep-wake routines.

Every session would separated by a 1-week interval. The average sleep duration (CON) is going to be estimated by using actigraphy Motionwatch 8 for 5 days (from Monday to Friday).

Female athletes will receive accelerometers one day before experimental sessions. Participants will be asked to wear them on their non-dominant wrists from 8 p.m. to the next morning (experimental sessions day).

The participants would complete the morning session with a battery of physical tests, measuring several components of specific physical performance capacity and cognitive function.

During the experimental sessions, participants would be at the luteal or follicular phases excluding the period of bleeding (4-5 days) and the time immediately before planned bleeding (3 days before), because this can have a bad influence on sleep.

ELIGIBILITY:
Inclusion Criteria:

* a minimum of 3 years of training experience;
* practicing physical activity for the last 6 months at least 3 times per week for 2h
* current medical qualification for competitive sport

Exclusion Criteria:

* diseases that can have a bad influence on the menstrual cycle (e.g. polycystic ovarian syndrome, endometriosis);
* using hormonal contraception;
* regularity of the menstrual cycle.
* diagnosed cardiovascular, metabolic, gastrointestinal, or neurological diseases;
* movement, neuromuscular or musculoskeletal disorders;
* taking medications and supplements that may affect fitness test results;
* taking supplements that may affect biochemical test results
* sleep disorders
* PSQI >5

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Maximal strength bench press test | 1 day after night with or without intervention
  The next day after a) sleep restriction b) normal sleep
Muscle endurance test in bench press | 1 day after night with or without intervention
  muscle endurance test in the bench press exercise at 50% 1RM
Explosive bench press exercise | 1 day after night with or without intervention
  three sets of three repetitions of explosive bench press exercise at 50% of the load representing one-repetition maximum (1RM)
Countermovement jump | 1 day after night with or without intervention
  Vertical jump test performed by having an athlete quickly squat to a self-selected depth and then jump as high as possible.

SECONDARY OUTCOMES:
Mood (POMS) | 1 day after night with or without intervention
  The POMS is a widely-applied measure for the assessment of an individual's mood. During each experimental session. Before sports performance protocol.
Pain (Pain scale) | 1 day after night with or without intervention
  A pain scale is a tool use to help assess a person's pain. Scale 0-10 (0- lack of pain; 10 - maximal pain). Immediately after the last performance exercise in experimental sessions.
Motivation | 1 day after night with or without intervention
  During each experimental session. Before sports performance protocol.
Rating perceived exertion (RPE) | 1 day after night with or without intervention
  A subjective scale that assesses the severity of effort exerted. Includes a rating from 6 perceiving "no effort" to 20 perceiving "maximum effort." Immediately after the last performance exercise in experimental sessions.
Stress and recovery (SRSS) | 1 day after night with or without intervention
  The Short Recovery and Stress Scale (SRSS) measure the recovery-stress state of an athlete multidimensionally with eight items on emotional, mental, physical, and overall levels. In the morning, each experimental day and the day after.
Readiness-to-train questionnaire (RTT-Q) | 1 day after night with or without intervention
  Subjective reactions related to the level of motivation for effort. In the morning, each experimental day and the day after.

OTHER OUTCOMES:
Objective Sleep - Total sleep time | 1 day after night with or without intervention
  Total sleep time obtained from sleep onset to time at wake-up assessed by actigraphy. The night before and after the experimental sessions.
Objective Sleep - Sleep efficiency | 1 day after night with or without intervention.
  The percentage of total sleep time to lights off and leaving bed assessed by actigraphy. The night before and after the experimental sessions.
Objective Sleep - WASO (Wake After Sleep Onset) | 1 day after night with or without intervention.
  The total number of minutes that a person is awake after having initially fallen asleep assessed by actigraphy. The night before and after the experimental sessions.
Objective Sleep - Sleep duration | 1 day after night with or without intervention.
  The quantity of time that a person sleeps assessed by actigraphy. The night before and after the experimental sessions.
Objective Sleep - Sleep onset time | 1 day after night with or without intervention.
  The time it takes a person to fall asleep after turning the lights out assessed by actigraphy. The night before and after the experimental sessions.
Objective Sleep - Wake time | 1 day after night with or without intervention.
  The hours in the day that a person is awake assessed by actigraphy. The night before and after the experimental sessions.
Blood collection - progesterone | 1 day after night with or without intervention.
  Blood will be drawn to measure progesterone. Before each experimental sesion
Blood collection - estradiol | 1 day after night with or without intervention.
  Blood will be drawn to measure estradiol. Before each experimental sesion

CONTACTS AND LOCATIONS:
Locations (1):
- University School of Physical Education in Cracow, Krakow, Poland